CLINICAL TRIAL: NCT00709631
Title: Prospective Evaluation of the Interest of a Systematic Biopsy for Hard-to-heal Leg Ulcers
Brief Title: Interest of a Systematic Biopsy for Hard-to-heal Leg Ulcers
Acronym: ULCERE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Other Study IDs: 00006477
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Leg Ulcers
Keywords: Malignant transformation of leg ulcer; MARJOLIN's ulcer; Biopsy; Leg ulcer; Chronic wound; Squamous cell carcinoma; Basal cell carcinoma
MeSH Terms: conditions — Leg Ulcer; Carcinoma, Squamous Cell; Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary aim of the study : to evaluate the prevalence of ulcerated cutaneous carcinoma or malignant degeneration, in leg ulcers, presumed of vascular origin and without evidence of healing despite 3 months of adequate treatmentSecondary aims of the study : to evaluate the interest of immunostainings for desmogleins 1-2 and p16 on biopsies to differentiate between pseudo epitheliomatous hyperplasia and squamous cell carcinoma ; and the prognosis of diagnosed carcinomas at 12 monthsStudy hypothesis : systematic biopsies of hard-to-heal leg ulcer may help to detect ulcerated carcinomas misdiagnosed as vascular ulcer or malignant degeneration of leg ulcer.

DETAILED DESCRIPTION:
Prospective multicentric inclusion of 150 patients with leg ulcers without any evidence of healing (no change or increase of ulcer area) despite 3 months of adequate treatment The study population consisted of consecutive patients with one or more leg ulcers, diagnosed as related to venous insufficiency, associated or not with concomitant arterial insufficiency. All patients undergo a standard treatment including compression therapy adapted to the ankle brachial index and a local treatment depending on the wound stage.At inclusion, systematic punch biopsies (5-6 mm) are taken as part of routine clinical care under local anaesthetic by an experienced clinician: 1 to 2 biopsies in the edges and 1 to 2 biopsies in the wound bedSpecimens are transported in formalin solution to the usual pathology laboratory of the investigator. At the end of the study, specimens will be sent for immunostainings in a single pathology laboratory (Rouen, France)Treatments and/or other investigations are decided by the investigatorAt 12 months of usual follow-up, final diagnosis and prognosis are noted in the study file by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* leg ulcer of more than 3 months of duration
* leg ulcer presumed of vascular origin
* adequate etiologic treatment since 3 months
* absence of evidence of healing : absence of reduction of wound area or increase in wound area and/or in depth

Exclusion Criteria:

* hypertensive ulcer
* vasculitis
* treatment by cytotoxic agents or steroids in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with one or more leg ulcers, diagnosed as related to venous insufficiency, associated or not with concomitant arterial insufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia SENET, MD, Principal Investigator — AP-HP, Hôpital Charles Foix, 94205 Ivry/Seine, France et Hôpital Tenon, 75020 Paris, France
Locations (1):
- Patricia SENET, MD, Ivry-sur-Seine, Île-de-France Region, France

REFERENCES:
- [Derived] Senet P, Combemale P, Debure C, Baudot N, Machet L, Aout M, Vicaut E, Lok C; Angio-Dermatology Group Of The French Society Of Dermatology. Malignancy and chronic leg ulcers: the value of systematic wound biopsies: a prospective, multicenter, cross-sectional study. Arch Dermatol. 2012 Jun;148(6):704-8. doi: 10.1001/archdermatol.2011.3362. PMID 22772403